CLINICAL TRIAL: NCT01457508
Title: Study to Assess the Immunogenicity and Reactogenicity of DTPa-HBV-IPV Vaccine Mixed With Hib Vaccine to Healthy Infants at 3, 5 and 11 Months of Age, Compared to Each Vaccine Administered Separately
Brief Title: Immunogenicity and Reactogenicity of DTPa-HBV-IPV/Hib, Compared to DTPa-HBV-IPV and Hib Administered Separately
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217744/054
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B; Diphtheria; Haemophilus Influenzae Type b (Hib); Poliomyelitis; Pertussis; Tetanus
Keywords: combination vaccine; DTPa-HBV-IPV; Hib
MeSH Terms: conditions — Hepatitis B; Diphtheria; Haemophilus Infections; Poliomyelitis; Whooping Cough; Tetanus | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Hiberix

ARMS (2):
- Group A (Experimental): Subjects will receive one single injection of DTPa-HBV-IPV vaccine mixed with Hib vaccine.
  Interventions: Biological: DTPa-HBV-IPV/Hib (Infanrix hexa™)
- Group B (Active Comparator): Subjects will receive two separate injections of DTPa-HBV-IPV and Hib vaccine.
  Interventions: Biological: DTPa-HBV-IPV (Infanrix penta™); Biological: Hib (Hiberix™)

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib (Infanrix hexa™) — Three doses administered intramuscularly
  Arms: Group A
Biological: DTPa-HBV-IPV (Infanrix penta™) — Three doses administered intramuscularly
  Arms: Group B
Biological: Hib (Hiberix™) — Three doses administered intramuscularly
  Arms: Group B

SUMMARY:
This study will assess the immunogenicity and safety of GlaxoSmithKline (GSK) Biologicals' (formerly SB Biologicals') DTPa-HBV-IPV/Hib (Infanrix hexa™) vaccine compared with separate administration of DTPa-HBV-IPV (Infanrix penta™) and Hib (Hiberix™) vaccine administered at 3, 5 and 11 (or 12) months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 3 months of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents or guardians of the subject after they have been advised of the risks and benefits of the study in a language which they clearly understood, and before performance of any study procedure.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply at the time of study entry, the subject must not be included in the study:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of chronic immunosuppressants or other immune-modifying drugs within three months before vaccination.
* Administration of a vaccine not foreseen by the study within 30 days before each dose of the study vaccines and ending 30 days after.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib disease.
* History of /or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio and/or Hib disease or infection.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including allergic reactions to neomycin and polymyxin B.
* Major congenital defects or serious chronic illness.
* History of seizures or of any neurological disease at study entry.
* Administration of immunoglobulins and/or any blood products since birth, or planned administration during the study period.
* Acute disease at time of enrolment

Ages: 12 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 1999-01; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccine in terms of number of subjects with antibody titres greater than or equal to cut off value | One month after the 2nd dose of the primary vaccination course ( Month 3)

SECONDARY OUTCOMES:
Immunogenicity with respect to the components of the study vaccines in terms of number of seroprotected subjects | One month after the 2nd dose ( Month 3), before and one month after the 3rd dose of the primary vaccination course ( Month 8 and 9)
Immunogenicity with respect to the components of the study vaccines in terms of number of seropositive subjects | One month after the 2nd dose ( Month 3), before and one month after the 3rd dose of the primary vaccination course ( Month 8 and 9)
Immunogenicity with respect to the components of the study vaccines in terms of antibody titres | One month after the 2nd dose ( Month 3), before and one month after the 3rd dose of the primary vaccination course ( Month 8 and 9)
Immunogenicity with respect to the components of the study vaccines in terms of vaccine response | One month after the 3rd dose ( Month 9), and one month after the 2nd dose of the primary vaccination course ( Month3)
Occurrence of solicited local symptoms | Within 4 days after each vaccination and overall
Occurrence of solicited general symptoms | Within 4 days after each vaccination and overall
Occurrence of unsolicited symptoms | Within 30 days after each vaccination and overall
Occurrence of serious adverse events | Throughout the entire study up to and including 30 days post-vaccination ( Month 0 to Month 9)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Crovari P. et al. Immunogenicity and reactogenicity of combined DTPa-HBV-IPV/Hib vaccine compared to concomitant administered DTPa-HBV-IPV and Hib vaccines given at 3, 5 and 11 months of age. Abstract presented at the 19th Annual Meeting ESPID, Istanbul, Turkey, 26-28 March 2001.
- [Background] Gabutti G, Zepp F, Schuerman L, Dentico P, Bamfi F, Soncini R, Habermehl P, Knuf M, Crovari P; Cooperative Italian Group for the Study of Combined Vaccines. Evaluation of the immunogenicity and reactogenicity of a DTPa-HBV-IPV Combination vaccine co-administered with a Hib conjugate vaccine either as a single injection of a hexavalent combination or as two separate injections at 3, 5 and 11 months of age. Scand J Infect Dis. 2004;36(8):585-92. doi: 10.1080/00365540410017572. PMID 15370670
- [Derived] Van Der Meeren O, Kuriyakose S, Kolhe D, Hardt K. Immunogenicity of Infanrix hexa administered at 3, 5 and 11 months of age. Vaccine. 2012 Apr 5;30(17):2710-4. doi: 10.1016/j.vaccine.2012.02.024. Epub 2012 Feb 18. PMID 22349525